CLINICAL TRIAL: NCT05970315
Title: Priorities Aligned Deprescribing for Persons Living With Dementia and Their Caregiver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Aanand Dinkar Naik, Professor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSC-SPH-22-0639; 5R24AG064025-05 (NIH)
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPC (Experimental)
  Interventions: Behavioral: PPC
- Usual Care (Active Comparator)
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: PPC — Participants will have an encounter with a facilitator who will identify priorities (outcome goals and care preferences) from the dyads and transmits them in the electronic health records (EHR), and a follow-up encounter with their usual geriatric care provider to decide upon changes in their care that align with the identified priorities.
  Arms: PPC
Behavioral: Usual care — Participants will have a geriatric clinic visit with a geriatrician that acts as their primary care provider (PCP) , in which the dyads will be encouraged by an unblinded study coordinator to ask about reducing medication burden.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to compare patient priorities care (PPC) and usual care (UC) patients to identify differences in post-encounter medication changes, treatment burden (TBQ), and shared decision making in Older Patient Assessment of Chronic Illness Care (OPACIC), to understand PPC participant's sense-making and communication approaches related to deprescribing decisions in relation to the identified health priorities and to identify and categorize adverse drug withdrawal events (ADWEs)

ELIGIBILITY:
Inclusion Criteria:

* Dementia listed as an active problem in the medical record, including Alzheimer's disease, vascular dementia, frontotemporal dementia, Parkinson's dementia, Lewy body disease.
* The functional assessment staging tool (FAST) score of 5 or lower (This will be established by the patient's clinician).
* 2 or more additional chronic conditions
* Takes 5 or more regular medications and
* A caregiver present during visits. Caregivers may include family members or unrelated caregivers and will be identified through chart review and confirmed by clinician, patient, and surrogate decision maker if necessary. Identified caregivers must be involved in decisions and care of People living with dementia (PLWD) and routinely attend clinic visits with patient

Exclusion Criteria:

* FAST score of 6 or more (This will be established by the patient's clinician).
* Significant hearing, vision, or advanced cognitive impairment that limits ability to participate in PPC encounters,
* Caregiver is unwilling or able to participate in visits, or
* Deemed ineligible by their Primary care physician (PCP)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Number of medication changes | Baseline, 3 month
Type of medication changes | Baseline, 3 month
Change in patient reported treatment burden as assessed by the Treatment Burden Questionnaire (TBQ) | Baseline, 3 month
  This is a 15 item questionnaire and each is scored from 0(not a problem) to 10(big problem) for a maximum score of 150, higher number indicating more burden
Number, likelihood, and severity of adverse drug reactions (ADRs) as assessed by the Naranjo scale | 3 months
  Naranjo scale is a 10 item questionnaire.Total scores range from -4 to +13; the reaction is considered definite if the score is 9 or higher, probable if 5 to 8, possible if 1 to 4, and doubtful if 0 or less.
Number, likelihood, and severity of adverse drug withdrawal events (ADWEs) as assessed by the Naranjo scale | 3 months
  Naranjo scale is a 10 item questionnaire.Total scores range from -4 to +13; the reaction is considered definite if the score is 9 or higher, probable if 5 to 8, possible if 1 to 4, and doubtful if 0 or less.

SECONDARY OUTCOMES:
Patient perceived chronic disease care as assessed by the Older Patient Assessment of Chronic Illness Care (OPACIC) score | Baseline, 3 months
  This is a 10 item questionnaire and each is scored from 1(almost never) to 5(almost always),for a maximum score of 50 ,higher scores indicate better perceived chronic disease care

CONTACTS AND LOCATIONS:
Overall Officials: Aanand D Naik, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No